CLINICAL TRIAL: NCT00855413
Title: CID 0821 - Pilot Study to Evaluate HIV Viremia and Persistence in Acutely HIV-Infected Antiretroviral Naïve Patients Treated With Darunavir/Ritonavir and Etravirine
Brief Title: HIV Viremia and Persistence in Acutely HIV-Infected Patients Treated With Darunavir/Ritonavir and Etravirine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted by sponsor due to slow enrollment.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Cynthia L Gay, MD, Clinical Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CID 0821
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-09

CONDITIONS: Acute HIV Infection; HIV Infections
Keywords: Acute HIV; HIV; Treatment Naive; Acute Infections
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Ritonavir; etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Darunavir/Ritonavir and Etravirine (Other): Darunavir/Ritonavir 800 mg/100 mg orally once daily.
  ETR will be given 200 mg orally twice daily, although patients may choose to take ETR 400 mg QD to have a simpler all QD regimen.
  Interventions: Drug: Darunavir; Drug: Ritonavir; Drug: Etravirine

INTERVENTIONS:
Drug: Darunavir — 800 mg orally once daily
  Other Names: Prezista
Drug: Ritonavir — 100 mg orally once daily
  Other Names: Norvir
Drug: Etravirine — 200 mg orally twice daily, although patients may choose to take ETR 400 mg QD to have a simpler all QD regimen
  Other Names: Intelence

SUMMARY:
Purpose: This is a pilot study to evaluate HIV viremia and persistence in acutely HIV infected antiretroviral naïve patients treated with Darunavir/ritonavir and Etravirine

Participants: 20 participants, age 18 and older, HIV infected, antiretroviral naïve patients

Procedures (methods): ARV treatment with Darunavir/ritonavir and Etravirine,

Optional studies:

Genital secretion samples, Cerebrospinal fluid samples, Leukapheresis, Endoscopy/colonoscopy

DETAILED DESCRIPTION:
Study Design

This is a multicenter, single arm, 48-week open-label pilot study of DRV/R & ETR in acute HIV infection. Study sites will be members of the Duke-UNC Acute HIV Infection Study Consortium. If baseline resistance is detected after treatment begins (e.g. evidence of pre-existing baseline resistance (genotypic or phenotypic) that may adversely affect the efficacy of the study regimen), the patient may elect to alter treatment as per best clinical practice. The new regimen will not be provided by the study, but will be obtained for the participant through available clinical resources.

After patients are identified with acute HIV infection, they will be offered the opportunity to participate in the study. Patients will also be offered the opportunity to co-enroll in CHAVI 001 and 012, studies that follow the virological and immunological response of patients with AHI, regardless of the initiation of ART. An overall consent form will be signed for study participation, and separate informed consents with signatures will be obtained for optional studies. Patients will be eligible for participation after signing the overall consent - agreeing to participate in studies of other compartment specimens is not required for enrollment. At the initial visit, patient eligibility will be confirmed with appropriate laboratory testing (see "STUDY POPULATION"). When eligibility is verified, entry laboratory studies will be obtained, and the participants will be started on DRV/r, and ETR. All participants will be followed at regular intervals thereafter as specified in the schedule of evaluations. Participants meeting criteria for virologic failure will be offered the opportunity to switch to the best available regimen as selected by their HIV provider.

Hypothesis

Combination therapy with DRV/R & ETR will suppress plasma viremia and improve immunologic function in antiretroviral (ART)-naïve, acutely HIV-infected (AHI) patients, and will limit replication in HIV-1 cellular compartments.

ELIGIBILITY:
Inclusion Criteria:

1. Documentation of Acute HIV Infection as defined above.
2. Men and women age ≥18 years.
3. Participants will be ART naïve, defined as ≤14 days of antiretroviral treatment at any time prior to entry. The only exceptions are: Post-exposure prophylaxis (PEP) provided the patient was documented as HIV-1 negative at least 3-6 months after completion of the PEP treatment.
4. Screening HIV-1 RNA >1,000 copies/mL obtained within 30 days at study entry.
5. Lab values obtained within 30 days prior to study entry:
6. Absolute neutrophil count >500/mm3
7. Hemoglobin > 8.5 g/dL for men and > 8.0 g/dL for women
8. Platelet count >50,000/mm3
9. AST (SGOT) ≤2.5 x ULN
10. ALT (SGPT) ≤2.5 x ULN
11. Total bilirubin <2.5 x ULN
12. Calculated creatinine clearance (Cockcroft-Gault formula) > 30mL/min:

    * CrCl = (140-age) x body weight (kg) (x 0.85 if female)
    * Serum creatinine [mg/dL] x (72)
13. For women of reproductive potential, a negative serum or urine pregnancy test within 7 days prior to initiating antiretroviral study medications. Reproductive potential is defined as females who have reached menarche and have not been post-menopausal for at least 24 consecutive months, or have not undergone surgical sterilization (e.g., hysterectomy, bilateral oophorectomy, or salpingotomy). Acceptable documentation of surgical sterilization includes patient-reported history.
14. If participating in sexual activity that could lead to pregnancy, female study patients must use at least one form of contraception, which could consist only of a barrier method. All patients must continue to use contraception for 6 weeks after stopping the study medications. Acceptable methods of contraception include: condoms (male or female) with or without spermicidal agent, diaphragm or cervical cap with spermicide, or IUD. Female volunteers not of reproductive potential are not required to use contraception.
15. Ability and willingness of patient to give written informed consent.

Exclusion Criteria:

1. Women who are pregnant or breast-feeding.
2. Women with a positive pregnancy test on enrollment or prior to study drug administration.
3. Women of reproductive potential who are unwilling or unable to use acceptable methods to avoid pregnancy for the entire study period
4. Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry.

   * Prednisone at a daily dose of 10 mg or less (physiologic replacement dose) is permitted.
5. Known allergy/sensitivity to study drugs or their formulations.
6. Difficulty swallowing capsules/tablets.
7. Inability to communicate effectively with study personnel.
8. Incarceration; prisoner recruitment and participation are not permitted.
9. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements or confound the analysis of study endpoints.
10. Any active psychiatric illness including schizophrenia, severe depression, or severe bipolar affective disorder that, in the opinion of the investigator, could confound the analysis of the neurological examination or neuropsychological test results.
11. Active brain infection (except for HIV-1), brain neoplasm, space-occupying brain lesion requiring acute or chronic therapy. Participants with any fungal meningitis, parasitic infection, or CNS lymphoma are excluded from participation.
12. Serious illness requiring systemic treatment and/or hospitalization until patient either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 7 days prior to study entry. NOTE: Oral candidiasis, vaginal candidiasis, mucocutaneous herpes simplex, and other minor illnesses (as judged by the site investigator) have no restriction.
13. Known cardiac conduction disease.
14. Prior treatment with any other experimental drug for any indication (within 30 days of initiating study treatment).
15. Unable to discontinue any current medications that are excluded during study treatment.
16. A life expectancy less than twelve months.
17. Acute Viral Hepatitis, including, but not limited to, Hepatitis A, B, or C
18. Chronic Hepatitis B Infection documented by a detectable serum Hepatitis B surface antigen (HBsAg) or plasma HBV DNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Gay, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; David M Margolis, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - The University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina

REFERENCES:
- [Background] Gay CL, Mayo AJ, Mfalila CK, Chu H, Barry AC, Kuruc JD, McGee KS, Kerkau M, Sebastian J, Fiscus SA, Margolis DM, Hicks CB, Ferrari G, Eron JJ; Duke-UNC Acute HIV Infection Consortium. Efficacy of NNRTI-based antiretroviral therapy initiated during acute HIV infection. AIDS. 2011 Apr 24;25(7):941-9. doi: 10.1097/QAD.0b013e3283463c07. PMID 21487250
- [Background] C Gay, O Dibben, A Stacey, N Gasper-Smith, M Liu, N Goonetilleke, G Ferrari, J Eron, C Hicks, A McMichael, B Haynes, P Borrow, M Cohen, the Duke-UNC CHAVI 001 Clinical Working Group. "Effect(s) of antiretroviral treatment on acute HIV infection." XVII International AIDS Conference, 2008 Abstract no. THPE0086.
- [Derived] Gay CL, Neo DT, Devanathan AS, Kuruc JD, McGee KS, Schmitz JL, Sebastian J, Shaheen NJ, Ferrari G, McKellar M, Fiscus SA, Hicks CB, Robertson K, Kashuba ADM, Eron JJ, Margolis DM. Efficacy, pharmacokinetics and neurocognitive performance of dual, NRTI-sparing antiretroviral therapy in acute HIV-infection. AIDS. 2020 Nov 1;34(13):1923-1931. doi: 10.1097/QAD.0000000000002652. PMID 32773474

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals diagnosed with acute HIV in clinical sites within 30 days of enrollment and at least 18 years of age were enrolled. Acute HIV defined as: i) negative EIA and positive NAT; ii) positive EIA and positive NAT with negative/indeterminate western blot (WB); or iii) positive EIA, positive WB and EIA negative documentation in prior 30 days.
Groups:
- Acute HIV Infection Treatment Group: All participants were administered darunavir 800mg, ritonavir 100mg once daily plus etravirine as 400mg once daily or 200mg twice daily started within 30 days of acute HIV diagnosis and continued for 48 weeks. Participants were evaluated on study at weeks 2, 4, 8, 12, 16, 24 and 48.
Period: Overall Study
Arm/Group | Acute HIV Infection Treatment Group
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] — Median age and range of all participants enrolled in study Population: years
  years
    Age | 23 [19 to 51]
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of participants enrolled onto the study
  Participants
    Female | 2
    Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Region of enrollment for all participants
  participants
    United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Virologic Response
Description: Virologic response defined as plasma HIV RNA measurement <200 copies/mL at week 24
Time Frame: 24 weeks
Population: All participants enrolled were included in analysis of virologic response
Measure: Count of Participants; unit: Participants
Groups:
- Acute HIV Infection Treatment Group: Participants received darunavir 800mg, ritonavir 100mg once daily plus etravirine as 400mg once daily or 200mg twice daily started within 30 days of acute HIV diagnosis.
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 15
Participants | 13

2. Secondary Outcome: Number of Participants With Virologic Response
Description: Virologic response to study treatment defined as plasma HIV RNA measurement <50 copies/mL at week 48
Time Frame: 48 weeks from enrollment
Population: All participants retained on study through week 48 were included in the analysis of virologic efficacy at week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 12
Participants | 9

3. Secondary Outcome: Median Change in CD4 Cell Count From Week 0 to Week 24.
Time Frame: week 0, week 24
Population: All participants enrolled were included in this analysis
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 15
cells/mm^3 | 158 [-281 to 916]

4. Secondary Outcome: Median Change in CD4 Cell Count From Week 0 to Week 48.
Time Frame: 48 weeks from enrollment
Population: 12 participants with a week 48 study visit were included in analysis
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 12
cells/mm^3 | 349 [7 to 495]

5. Secondary Outcome: HIV RNA Levels Immediately Prior to Initiating Study Treatment.
Time Frame: HIV RNA level at enrollment
Measure: Median (Full Range); unit: copies/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 15
copies/mL | 1,000,000 [22,858 to 29,807,640]

6. Secondary Outcome: Median Time to HIV RNA Suppression to <200 Copies/mL
Time Frame: From enrollment to the date of HIV RNA suppression, assessed up to Week 48
Measure: Median (Full Range); unit: days
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 15
days | 59 [15 to 187]

7. Secondary Outcome: HIV RNA Detection in Semen
Description: Total cumulative levels of HIV RNA detected in the semen of participants from enrollment through week 48.
Time Frame: From enrollment through 48 weeks
Population: Study stopped prior to target enrollment by sponsor. Given insufficient semen samples, correlation of HIV viremia in semen with time to suppression was not performed due to inadequate power to analyze the outcome.
Measure: Mean (Full Range); unit: copies/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
copies/mL | 2541 [0 to 7470]

8. Secondary Outcome: Number of Participants Who Stopped Study Treatment Due to Adverse Event or Intolerance
Time Frame: Enrollment to Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 15
Participants | 1

9. Secondary Outcome: Adverse Events Possibly or Definitely Related to Study Treatment Through Week 48
Description: Total number of adverse events observed that were possibly or definitely related to study treatment through week 48
Time Frame: Enrollment to week 48
Measure: Number; unit: adverse events
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 15
adverse events | 13

10. Secondary Outcome: Maximum Etravirine Exposure in Cerebrospinal Fluid Among Participants Who Consented to an Optional Lumbar Puncture
Time Frame: Week 4 and week 48
Population: 4 participants consented to 7 optional lumbar punctures to provide CSF samples for measurement of drug levels.
Measure: Number; unit: ng/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
ng/mL | 25

11. Secondary Outcome: Minimum Etravirine Exposure in Cerebrospinal Fluid Among Participants Who Consented to an Optional Lumbar Puncture
Time Frame: Week 4 and week 48
Population: 4 participants consented to 7 optional lumbar puncture to provide CSF sample for measurement of drug levels.
Measure: Number; unit: ng/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
ng/mL | 4

12. Secondary Outcome: Maximum Darunavir Exposure in Cerebrospinal Fluid Among Participants Who Consented to an Optional Lumbar Puncture
Time Frame: Week 4 and week 48
Population: Four participants consented to 7 optional lumbar puncture to provide CSF sample for measurement of drug levels.
Measure: Number; unit: ng/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
ng/mL | 240

13. Secondary Outcome: Minimum Darunavir Exposure in Cerebrospinal Fluid Among Participants Who Consented to an Optional Lumbar Puncture
Time Frame: Week 4 and week 48
Population: Four participants consented to 7 optional lumbar puncture to provide CSF sample for measurement of drug levels.
Measure: Number; unit: ng/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
ng/mL | 10

14. Secondary Outcome: Maximum Ritonavir Exposure in Cerebrospinal Fluid Among Participants Who Consented to an Optional Lumbar Puncture
Time Frame: Week 4 and Week 48
Population: Four participants consented to 7 optional lumbar puncture to provide CSF sample for measurement of drug levels.
Measure: Number; unit: ng/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
ng/mL | 22

15. Secondary Outcome: Minimum Ritonavir Exposure Range in Cerebrospinal Fluid Among Participants Who Consented to an Optional Lumbar Puncture
Time Frame: Week 4 and week 48
Population: Four participants consented to 7 optional lumbar puncture to provide CSF sample for measurement of drug levels.
Measure: Number; unit: ng/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
ng/mL | 2

16. Secondary Outcome: Maximum Etravirine Exposure in Semen Among Participants Who Consented to an Optional Collection of Semen
Time Frame: Weeks 0-4 and weeks 12, 48
Population: Four participants consented to provide a semen sample for measurement of drug levels.
Measure: Number; unit: ng/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
ng/mL | 185

17. Secondary Outcome: Minimum Etravirine Exposure in Semen Among Participants Who Consented to an Optional Collection of Semen
Time Frame: Weeks 0-4 and weeks 12, 48
Population: Four participants consented to provide a semen sample for measurement of drug levels.
Measure: Number; unit: ng/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
ng/mL | 12

18. Secondary Outcome: Maximum Darunavir Exposure in Semen Among Participants Who Consented to an Optional Collection of Semen
Time Frame: Weeks 0-4 and weeks 12, 48
Population: Four participants consented to provide a semen sample for measurement of drug levels.
Measure: Number; unit: ng/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
ng/mL | 1296

19. Secondary Outcome: Minimum Darunavir Exposure Range in Semen Among Participants Who Consented to an Optional Collection of Semen
Time Frame: Weeks 0-4 and weeks 12, 48
Population: Four participants consented to provide a semen sample for measurement of drug levels.
Measure: Number; unit: ng/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
ng/mL | 9

20. Secondary Outcome: Maximum Ritonavir Exposure in Semen Among Participants Who Consented to an Optional Collection of Semen
Time Frame: Weeks 0-4 and Weeks 12, 48
Population: Four participants consented to provide a semen sample for measurement of drug levels.
Measure: Number; unit: ng/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
ng/mL | 22

21. Secondary Outcome: Minimum Ritonavir Exposure in Semen Among Participants Who Consented to an Optional Collection of Semen
Time Frame: Weeks 0-4 and Weeks 12, 48
Population: Four participants consented to provide a semen sample for measurement of drug levels.
Measure: Number; unit: ng/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
ng/mL | 2

22. Secondary Outcome: Maximum Etravirine Exposure in Ileal Tissue Among Participants Who Consented to an Optional Gut Biopsy Procedure
Time Frame: between Week 4-12 and between Weeks 36-48
Population: Six participants consented to ileal biopsy for measurement of drug levels
Measure: Number; unit: ng/g
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 6
ng/g | 83,749

23. Secondary Outcome: Minimum Etravirine Exposure Range in Ileal Tissue Among Participants Who Consented to an Optional Gut Biopsy Procedure
Time Frame: between Week 4-12 and between Weeks 36-48
Population: Six participants consented to ileal biopsy for measurement of drug levels
Measure: Number; unit: ng/g
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 6
ng/g | 34

24. Secondary Outcome: Maximum Darunavir Exposure Range in Ileal Tissue Among Participants Who Consented to an Optional Gut Biopsy Procedure
Time Frame: between Week 4-12 and between Weeks 36-48
Population: Six participants consented to ileal biopsy for measurement of drug levels
Measure: Number; unit: ng/g
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 6
ng/g | 83,749

25. Secondary Outcome: Minimum Darunavir Exposure Range in Ileal Tissue Among Participants Who Consented to an Optional Gut Biopsy Procedure
Time Frame: between week 4-12 and between weeks 36-48
Population: Six participants consented to ileal biopsy for measurement of drug levels
Measure: Number; unit: ng/g
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 6
ng/g | 987

26. Secondary Outcome: Maximum Ritonavir Exposure Range in Ileal Tissue Among Participants Who Consented to an Optional Gut Biopsy Procedure
Time Frame: between week 4-12 and between Weeks 36-48
Population: Six participants consented to ileal biopsy for measurement of drug levels
Measure: Number; unit: ng/g
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 6
ng/g | 14,698

27. Secondary Outcome: Minimum Ritonavir Exposure Range in Ileal Tissue Among Participants Who Consented to an Optional Gut Biopsy Procedure
Time Frame: between week 4-12 and between weeks 36-48
Population: Six participants consented to ileal biopsy for measurement of drug levels
Measure: Number; unit: ng/g
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 6
ng/g | 96

28. Secondary Outcome: Number of Participants With HIV RNA Measurement Above the Limits of Detection in Cerebrospinal Fluid
Time Frame: Week 4 and Week 48
Population: Four participants provided 7 CSF samples for measurement of HIV RNA level
Measure: Number; unit: participants
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 4
participants | 0

29. Secondary Outcome: Number of Participants With Neurocognitive Impairment at Baseline
Time Frame: Week 2 or 4
Population: Participants who consented to optional procedure of neurocognitive assessment at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 13
Participants | 8

30. Secondary Outcome: Number of Participants With Neurocognitive Impairment at Week 24
Time Frame: Week 24
Population: Participants who consented to optional procedure of neurocognitive assessment at week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 9
Participants | 3

31. Secondary Outcome: Number of Participants With Neurocognitive Impairment at Week 48
Time Frame: Week 48
Population: Participants who consented to optional procedure of neurocognitive assessment at week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 10
Participants | 3

32. Secondary Outcome: Overall Neurocognitive Impairment Score at Week 2 or 4
Description: Neuropsychological performance was assessed at Week 2 or 4, Week 24 and Week 48 in the following measures: Premorbid/language (Wide Range Achievement Test 4 -Reading Subtest), Learning (HVLT-R, Hopkins Verbal Learning Test-Revised), Memory (HVLT-R), Speed of Processing (Trailmaking A (Army Individual Test Battery, 1944), 1974, Stroop color, Attention (WAIS-III Symbol Search; Stroop word, Fine motor, Executive (Trailmaking B, Stroop interference, Letter, Category Fluency. An overall summary score was created by averaging all tests. Participants also completed the self-reported functional status Patient's Assessment of Own Functioning Inventory (PAOFI) and the Activities of Daily Living Scale (ADLS). Best available demographically corrected normative data were utilized to create z scores. A negative z score denotes below-average performance relative to a US normative comparison population. A higher z score is a better outcome.
Time Frame: Week 2 or 4
Population: participants who underwent neurocognitive assessment at week 2 or 4
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 10
z score | -0.69 (.14)

33. Secondary Outcome: Overall Neurocognitive Impairment at Week 24
Description: Neuropsychological performance was assessed at week 2 or 4, week 24 and week 48 in the following measures: Premorbid/language (Wide Range Achievement Test 4 -Reading Subtest), Learning (Hopkins Verbal Learning Test - Revised), Memory (HVLT-R), Speed of Processing (Trailmaking A (Army Individual Test Battery, 1944), 1974, Stroop color, Attention (WAIS-III Symbol Search; Stroop word, Fine motor, Executive (Trailmaking B, Stroop interference, Letter, Category Fluency. An overall summary score of neurocognitive functioning was created by averaging all tests. Participants also completed Patient's Assessment of Own Functioning Inventory (PAOFI) and the Activities of Daily Living Scale (ADLS). Best available demographically corrected normative data were utilized to create z scores. A negative z score denotes below-average performance relative to a US normative comparison population. A higher z score is a better outcome.
Time Frame: Week 24
Population: participants who underwent neurocognitive assessment at baseline and week 24
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 9
z score | -0.40 (.15)

34. Secondary Outcome: Overall Neurocognitive Impairment at Week 48
Description: Neuropsychological performance was assessed at baseline (week 2 or 4), week 24 and week 48 in the following domain (measures): Premorbid/language (Wide Range Achievement Test (WRAT) 4 - Reading Subtest), Learning (HVLT-R, Hopkins Verbal Learning Test - Revised), Memory (HVLT-R), Speed of Processing (Trailmaking A (Army Individual Test Battery, 1944), 1974, Stroop color, Attention (WAIS-III Symbol Search; Stroop word, Fine motor, Executive (Trailmaking B, Stroop interference, Letter, Category Fluency. An overall summary score of neurocognitive functioning was created by averaging all tests. Participants also completed the self-reported functional status Patient's Assessment of Own Functioning Inventory (PAOFI) and the Activities of Daily Living Scale (ADLS). Best available demographically corrected normative data were utilized to create z scores. A negative z score denotes below-average performance relative to a US normative comparison population. A higher z score is a better outcome.
Time Frame: Week 48
Population: participants who underwent neurocognitive assessment at baseline and week 48
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 10
z score | -.45 (.15)

35. Secondary Outcome: Change in Overall Neurocognitive Impairment From Baseline to Week 24 or 48
Description: Change in overall z score from baseline to week 24 or 48. A negative z score denotes below-average performance relative to a US normative comparison population. A higher z score is a better outcome.
Time Frame: Baseline to Week 24 or 48
Population: Participants who underwent neurocognitive assessment at baseline and Week 24 and/or 48.
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 11
z score | 4.23 (.15)
Statistical Analysis 1: Comparison: Acute HIV Infection Treatment Group; An overall summary score of neurocognitive functioning was created by averaging all tests. Best available demographically corrected normative data were utilized to create z scores and then deficit scores for impairment ratings.Change in neurocognitive functioning was analyzed using a one sided repeated measures ANOVA with neurocognitive performance as the dependent variable (total z score) and time (visit) as the independent variable. Degrees of freedom were 2,17; Test type: Other — one sided ANOVA; p = 0.03, ANOVA — The degrees of freedom (df) for the within factor (number of visits - 1) was 2, and the second df is the error df of 17; Mean Difference (Final Values) = 4.23, Standard Deviation 0.15

36. Secondary Outcome: Correlation of HIV RNA Levels in CSF and Drug Levels With Neurocognitive Functioning
Time Frame: From enrollment through Week 48
Population: Participants who consented to neurocognitive assessments at baseline and week 24 or 48. Sponsor stopped study prior to target enrollment.
Measure: Number; unit: r value
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 11
r value | NA — Insufficient CSF samples which were all below detectible limits for HIV RNA assay resulted in insufficient power to assess for correlations

37. Secondary Outcome: Correlation of Time to HIV RNA Levels <200 Copies/mL With Improvement in Neurocognitive Functioning From Baseline to Week 24 and 48
Time Frame: Baseline to Week 24 and 48
Population: Participants who consented to optional neurocognitive assessments at baseline and week 24 or 48
Measure: Number; unit: r value
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 11
r value | -.82
Statistical Analysis 1: Comparison: Acute HIV Infection Treatment Group; Correlation between time (days) to HIV RNA suppression <200 copies/mL and total z score (mean) was assessed by Spearman correlation; Test type: Other — Spearman correlation; p < .005, Spearman correlation — R = -0.82; spearman correlation = -.82; Correlation between time (days) to HIV RNA suppression <200 copies/mL and total z score (mean) was assessed by Spearman correlation

38. Secondary Outcome: HIV RNA Detection in Ileal Biopsy Specimens
Description: Average HIV RNA detected in the ileal biopsy specimens per participant over weeks 4 and 48.
Time Frame: Weeks 4 and 48
Population: Study stopped prior to target enrollment by sponsor. Given insufficient ileal biopsy samples, correlation of HIV viremia in ileal biopsies with time to suppression was not performed due to inadequate power to analyze the outcome.
Measure: Mean (Full Range); unit: copies/mL
Arm/Group | Acute HIV Infection Treatment Group
Number analyzed (Participants) | 6
copies/mL | 40 [0 to 506]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant over the 96 weeks of the study.
Description: Adverse events were assessed at each visit and graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events.
Groups:
- Darunavir/Ritonavir and Etravirine: Darunavir/Ritonavir and Etravirine
  DRV/r will be administered 800 mg/100 mg orally once daily.
  ETR will be given 200 mg orally twice daily, although patients may choose to take ETR 400 mg QD to have a simpler all QD regimen.
  Darunavir/Ritonavir and Etravirine: DRV/r will be administered 800 mg/100 mg orally once daily.
  ETR will be given 200 mg orally twice daily, although patients may choose to take ETR 400 mg QD to have a simpler all QD regimen.
Arm/Group | Darunavir/Ritonavir and Etravirine
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darunavir/Ritonavir and Etravirine (N=15)
Blood Cholesterol Increased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination prior to target enrollment due to slow enrollment limited analysis involving optional procedures. Lack of paired (baseline and followup) samples from optional procedures also limited ability to perform these analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes